CLINICAL TRIAL: NCT00644917
Title: Clinical Evaluation of the Phototoxic Potential of Xenaderm Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: H. B. Slade, M.D., Healthpoint, Ltd.
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: 011 101 09 001
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: wound healing; phototoxicity; Healthy Subjects
MeSH Terms: conditions — Dermatitis, Phototoxic | interventions — Granulex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Drug
  Interventions: Drug: Xenaderm
- B (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo
- C (No Intervention): Subjects serve as own controls.

INTERVENTIONS:
Drug: Xenaderm — 20mg under Finn chambers
  Arms: A
Drug: Placebo — 20mg under Finn chambers
  Arms: B

SUMMARY:
The product is being tested to see if exposure to light causes toxic reactions on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Innes Cargill, PhD, Study Director — Healthpoint, Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 1 study was conducted at one investigational site (Research Laboratory) located in the US, and conducted on healthy adult subjects of either gender, and skin-type I, II, or III, who were 18 years of age and older, from 19-Feb-2008 to 29-Feb-2008.
Groups:
- Xenaderm Ointment - Subjects Acted as Own Comparator: Two 20 mg samples of Xenaderm Ointment and two 20 mg samples of Vehicle were applied in Finn Chambers to four test sites of the left side of each subject's back; a fifth test site was covered with an empty Finn Chamber as a control site
Period: Overall Study
Arm/Group | Xenaderm Ointment - Subjects Acted as Own Comparator
Started | 38
Completed | 36
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Xenaderm vs. Vehicle - Subjects Acted as Own Comparator: Subjects received duplicate 20 mg applications of Xenaderm Ointment and Xenaderm vehicle contained in Finn Chambers, to the left sides of their backs
Arm/Group | Xenaderm vs. Vehicle - Subjects Acted as Own Comparator
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Skin Reaction Score
Description: Scores for phototoxic skin irritation were used to evaluate safety. In this study, irritation was graded using a scale that ranged from 0 (no reaction) to 7 (large vesiculo-bullous reaction) in whole units.
Time Frame: 48 hours
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Xenaderm Ointment - Irradiated: 20 mg samples of Xenaderm Ointment applied in a Finn Chambers to test site the left side of each subject's back - then irradiated
- Xenaderm Vehicle - Irradiated: 20 mg sample of Vehicle applied in Finn Chamber to test site on the left side of each subject's back - then irradiated
- Control - Irradiated: test site was covered with an empty Finn Chamber as a control site - then irradiated
- Xenaderm Ointment - Non-irradiated: 20 mg samples of Xenaderm Ointment applied in a Finn Chambers to test site the left side of each subject's back - not irradiated
- Xenaderm Vehicle - Non-irradiated: 20 mg samples of Xenaderm Vehicle applied in a Finn Chambers to test site the left side of each subject's back - not irradiated
Arm/Group | Xenaderm Ointment - Irradiated | Xenaderm Vehicle - Irradiated | Control - Irradiated | Xenaderm Ointment - Non-irradiated | Xenaderm Vehicle - Non-irradiated
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36
units on a scale
  Day 2 at patch removal | 0.4 (0.5) | 0.5 (0.6) | 0.1 (0.2) | 0.4 (0.5) | 0.5 (0.6)
  Day 2 immediately post UV radiation | 0.3 (0.6) | 0.7 (0.9) | 0.5 (0.8) | 0.2 (0.5) | 0.4 (0.6)
  Day 3 - 24 hours post UV radiation | 0.5 (1.0) | 0.8 (1.1) | 0.9 (1.1) | 0.3 (0.6) | 0.2 (0.4)
  Day 4 - 48 hours post UV radiation | 0.4 (0.8) | 0.6 (1.0) | 0.7 (1.1) | 0.2 (0.5) | 0.2 (0.5)

ADVERSE EVENTS:
Time Frame: All subjects were exposed to Xenaderm Ointment and Xenaderm vehicle at Day 1. The exposures were occluded under Finn Chambers for 24 hours.
Description: Tabulations of adverse events were used to qualitatively summarize the events by description, severity, and causality. The tabulations were reviewed for evidence of safety trends unrelated to the phototoxicity assessments.
Arm/Group | Xenaderm Ointment - Subjects Acted as Own Comparator
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 3/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenaderm Ointment - Subjects Acted as Own Comparator (N=36)
Skin Irritation (Skin and subcutaneous tissue disorders) | 3 (3) — Tape Irritation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less